CLINICAL TRIAL: NCT07075237
Title: A Study on the Efficacy and Functional Recovery of Switching From Oral Antipsychotics to Paliperidone Palmitate Injection in the Treatment of Schizophrenia
Brief Title: Efficacy and Functional Recovery After Switching From Paliperidone Palmitate Injection to Oral Antipsychotics in Schizophrenia
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Jiangsu Province Nanjing Brain Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JiangsuPNBH
Record Dates: First submitted 2025-07-11; First posted 2025-07-20 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Paliperidone Palmitate; Oral antipsychotics; Social function|
MeSH Terms: conditions — Schizophrenia; Social Adjustment | interventions — Paliperidone Palmitate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment group (Experimental): Switching from Oral Antipsychotics to Paliperidone Palmitate Injection in the Treatment of Schizophrenia Patients
  Interventions: Drug: Paliperidone Palmitate Injection (PP1M)

INTERVENTIONS:
Drug: Paliperidone Palmitate Injection (PP1M) — Day 0: 150 mg deltoid injection; Day 7: 100 mg deltoid injection; Monthly maintenance dose of 75-150 mg (deltoid or gluteal) for 6 months (dose adjusted per investigator's judgment).
  To avoid missed doses, administration is permitted ±7 days around the scheduled monthly date.

SUMMARY:
To evaluate the efficacy of Paliperidone Palmitate Injection in replacing oral antipsychotics for the treatment of schizophrenia and its impact on social function

DETAILED DESCRIPTION:
This study plans to enroll 120 patients diagnosed with schizophrenia per DSM-5 criteria who have achieved clinical stability on oral antipsychotic therapy. Patients will receive monotherapy with Paliperidone Palmitate Injection. Assessments will be conducted at baseline, Day 35±7, Day 91±7, and Day 175±7. Adverse events and concomitant medications will be recorded during follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients or inpatients meeting DSM-5 diagnostic criteria forschizophrenia;
2. Aged 18-65 years (inclusive), regardless of gender;
3. Currently receiving first- or second-generation oral antipsychotics (excluding clozapine) with stable condition as assessed by the investigator, and PANSS total score ≤80 at screening and baseline;
4. Signed informed consent by the patient and/or guardian;

Exclusion Criteria:

1. Comorbid psychiatric diagnoses other than schizophrenia;
2. Severe physical diseases, intellectual disability, organic brain disorders, or mental disorders due to physical illnesses;
3. QTc interval >450 ms (male) or >460 ms (female);
4. History of psychoactive substance abuse (excluding tobacco) within the past 12 months, or significant suicidal/violent tendencies;
5. Current or history of tardive dyskinesia (TD), neuroleptic malignant syndrome (NMS), or severe extrapyramidal symptoms (EPS);
6. Treatment-resistant schizophrenia (failure of ≥2 adequate antipsychotic regimens of different compounds);
7. Hypersensitivity or inefficacy to risperidone or paliperidone; 8. Pregnancy, lactation, planned pregnancy, or failure to use effective contraception during the study;

9. Other conditions deemed unsuitable by the investigator. |

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
The Positive and Negative Syndrome Scale (PANSS) | Day 175±7
  The Positive and Negative Syndrome Scale (PANSS) is a standardized clinical assessment tool used to evaluate the severity of symptoms in patients with schizophrenia. It measures three domains:
  Positive Symptoms (e.g., hallucinations, delusions), Negative Symptoms (e.g., social withdrawal, blunted affect), General Psychopathology (e.g., anxiety, guilt). Scores are derived from a 30-item structured interview, with each item rated on a 7-point scale (1=absent to 7=extreme). Higher total scores indicate more severe symptomatology. Widely used in research and clinical settings, PANSS helps monitor treatment efficacy and disease progression.

SECONDARY OUTCOMES:
Personal and Social Performance (PSP) | Baseline, Day 35±7, Day 91±7, Day 175±7
  The Personal and Social Performance (PSP) scale is a clinician-rated assessment tool designed to measure an individual's social and personal functioning across four key domains: socially useful activities (e.g., work/studies), personal/social relationships, self-care, and disruptive/aggressive behaviors. Scores range from 0 to 100, with higher values indicating better functional capacity. Widely used in mental health research and clinical practice, it provides a standardized way to evaluate functional impairment and recovery progress in conditions like schizophrenia.
EuroQol-5 Dimensions (EQ-5D) | Baseline, Day 35±7, Day 91±7, Day 175±7
  The EQ-5D (EuroQol-5 Dimensions) is a standardized, self-reported questionnaire used to assess health-related quality of life. It evaluates five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, each rated across three or five severity levels (depending on the version: EQ-5D-3L or EQ-5D-5L). Widely applied in health economics and clinical research, it aids in cost-effectiveness analyses and treatment outcome comparisons.
Clinical Global Impression-Severity (CGI-S) | Baseline, Day 35±7, Day 91±7, Day 175±7
  A single-item, 7-point clinician rating (1=normal to 7=extremely severe) evaluating global psychiatric illness severity. Not diagnosis-specific, it provides rapid assessment of symptom intensity across mental disorders.
Extrapyramidal Symptom Rating Scale (SAS) | Baseline, Day 35±7, Day 91±7, Day 175±7
  A clinician-administered tool assessing drug-induced movement disorders, including parkinsonism, dystonia, and akathisia. Rates 10 items (e.g., rigidity, tremor) on a 0-4 severity scale (total range 0-40). Widely used to monitor antipsychotic side effects.
Barnes Akathisia Rating Scale (BARS) | Baseline, Day 35±7, Day 91±7, Day 175±7
  A structured scale measuring antipsychotic-induced akathisia (motor restlessness). Combines:
  Subjective distress (0-5) Objective movements (0-5) Global severity (0-5) Critical for differentiating akathisia from anxiety/agitation.
Abnormal Involuntary Movement Scale (AIMS) | Baseline, Day 35±7, Day 91±7, Day 175±7
  A 12-item observational tool screening tardive dyskinesia severity. Focuses on facial/oral, extremity, and truncal involuntary movements (rated 0-4 per item). Requires baseline/follow-up assessments for longitudinal monitoring.

OTHER OUTCOMES:
electrocardiogram (ECG) | Baseline, Day 35±7, Day 91±7, Day 175±7
  To analysis whether ECG QT Interval of participants show any significant trend with time changes.
Alanine Aminotransferase (ALT) | Baseline, Day 35±7, Day 91±7, Day 175±7
  To analysis whether ALT level of participants show any significant trend with time changes.
Glucose (GLU) | Baseline, Day 35±7, Day 91±7, Day 175±7
  To analysis whether GLU level of participants show any significant trend with time changes.
Total Cholesterol (TC) | Baseline, Day 35±7, Day 91±7, Day 175±7
  To analysis whether TC level of participants show any significant trend with time changes.
High-Density Lipoprotein Cholesterol (HDL-C) | Baseline, Day 35±7, Day 91±7, Day 175±7
  To analysis whether HDL-C level of participants show any significant trend with time changes.
Low-Density Lipoprotein Cholesterol (LDL-C) | Baseline, Day 35±7, Day 91±7, Day 175±7
  To analysis whether LDL-C level of participants show any significant trend with time changes.
Triglycerides (TG) | Baseline, Day 35±7, Day 91±7, Day 175±7
  To analysis whether TG level of participants show any significant trend with time changes.
Prolactin (PRL) | Baseline, Day 35±7, Day 91±7, Day 175±7
  To analysis whether PRL level of participants show any significant trend with time changes.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing Brain Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided